CLINICAL TRIAL: NCT00431483
Title: Clinical and Economic Impact of Interventions by a Clinical Pharmacist on Antibiotic Use on Surgical Wards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Alexandra Weber, Pharmacist, Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AW2007
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Bacterial Infections
Keywords: antibacterial agents; surgery; pharmacist; economics, pharmaceutical
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmaceutical counseling (Other)
  Interventions: Behavioral: pharmaceutical consulting

INTERVENTIONS:
Behavioral: pharmaceutical consulting — to measure if information and advice by a pharmacist has an impact on quality and quantity of prescribed antibacterials

SUMMARY:
The purpose of this study is to establish the impact of a pharmacist's recommendations regarding choice, dosing and duration of antibiotic therapy on quality and cost of antibiotic treatment on surgical wards.

DETAILED DESCRIPTION:
Inappropriate or incorrect use of antibacterials exerts selection pressure on pathogens potentiating emergence of resistance, puts patients at risk for unnecessary adverse drug reactions and potentially prolongs the length of stay in hospital thus increasing healthcare costs.

In an effort to improve the quality of antibiotic drug therapy on surgical wards of a large university hospital, specific consulting by a clinical pharmacist was established.

The objective of this study is to assess the impact of pharmaceutical consulting on the quality and costs of antibiotic use in surgical wards.

Comparison:

Within a control period the current pattern of antibiotic use is monitored. During the intervention period, the impact of the interventions made by the clinical pharmacist on antibiotic use is examined. One ward serves as a parallel control group; no intervention is being made on this ward throughout this study.

ELIGIBILITY:
Inclusion Criteria:

* female and male patients receiving antibiotics for a proven or suspected infection on designated surgical wards

Exclusion Criteria:

* patients under 18
* patients unable or unwilling to consent to their data being evaluated
* patients receiving antibiotics perioperatively as prophylaxis
* patients receiving antibiotics for less than 48hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
overall duration of antibiotic therapy during study period | Feb 2008

SECONDARY OUTCOMES:
iv to oral switch | Feb 2008
  number of courses of iv antibiotics switched to oral antibiotics; duration of iv treatment
compliance of treatment with hospital formulary for antibiotic therapy | Feb 2008
cost of antibiotic therapy | Feb 2008
number and duration of therapy with antibiotics with redundant spectra | Feb 2008

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Walter Jauch, Prof. Dr., Study Director — Klinikum Grosshadern
Locations (1):
- Luwig Maximilians University - Klinikum Grosshadern, Munich, Bavaria, Germany